CLINICAL TRIAL: NCT05490485
Title: Camrelizumab Plus Cisplatin in Advanced Cutaneous Squamous Cell Carcinoma: a Single-arm, Open, Single-center Phase II Study
Brief Title: Camrelizumab Combined With Cisplatin in the Treatment of Advanced Cutaneous Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Associate chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZCSCC-1
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-08

CONDITIONS: Squamous Cell Carcinoma of the Skin
MeSH Terms: interventions — camrelizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab (Experimental): Camrelizumab (PD-1 MAB) combined with cisplatin for advanced cutaneous squamous cell carcinoma
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab combined with cisplatin for advanced cutaneous squamous cell carcinoma
  Other Names: cisplatin

SUMMARY:
This study is a card Rayleigh bead single combined cisplatin treatment of advanced squamous cell carcinoma of the skin resistance of single arm phase II study, open, single center, plan in two years into the group of 20 cases with histologic diagnosis of lymph node metastasis or distant metastasis CSCC of (1) or surgery can't/couldn't thorough radiotherapy, CSCC of locally advanced (class 2), To evaluate the efficacy of camrelizumab (PD-1 mab) combined with cisplatin in the treatment of advanced CSCC.

DETAILED DESCRIPTION:
This study is a card Rayleigh bead single combined cisplatin treatment of advanced squamous cell carcinoma of the skin resistance of single arm phase II study, open, single center, plan in two years into the group of 20 cases with histologic diagnosis of lymph node metastasis or distant metastasis CSCC of (1) or surgery can't/couldn't thorough radiotherapy, CSCC of locally advanced (class 2), To evaluate the efficacy, safety and quality of life of patients with advanced CSCC treated with camrelizumab (PD-1 mab) combined with cisplatin.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years;
2. The ECOG score is 0-1, and the ECOG score of amputation patients can be widened to 2, indicating good organ function;
3. Histologically determined CSCC with lymph node metastases or distal metastases (class 1) or locally advanced CSCC inoperable/unable to undergo radical radiotherapy (class 2).
4. Measurable tumor lesions were assessed by ultrasonography or CT within 21 days before enrollment;
5. Estimated survival time ≥3 months.
6. Primary tumor site Description: squamous cell carcinoma with primary labial mucosa can be included. Patients with primary SCC in the anogenital region (large and small labia, penis, scrotum, and perianal region) were excluded. The primary site was the nose, and patients were enrolled only if the investigator could definitively identify the primary site as the skin and not the nasal mucosa extending outward into the skin.
7. Category 2 only: Cases in which the investigator considers surgery inappropriate include: 1. Recurrent CSCC at the same location after two or more surgical operations and unable to undergo radical resection; 2. Local infiltration of CSCC made complete resection impossible; 3. The location of CSCC lesions is special and the operation is difficult, which may lead to severe defects or dysfunction (such as removing all or part of the facial structure, nose or eye, or requiring amputation); 4. Cases that are not suitable for surgical treatment for other reasons.
8. Category 2 only: At least one of the following criteria must be met if the investigator deems radiotherapy inappropriate: 1. The subject has received CSCC radiation therapy such that further radiation therapy would exceed the threshold for acceptable cumulative dose; 2. Subjects were intolerant to radiotherapy; 3. The subject is unwilling to participate in radiotherapy; 4. Cases in which radiotherapy is not suitable for other reasons.
9. Tumor histology: Patients with mixed histology (e.g., sarcomatoid carcinoma, adenosquamous carcinoma) are generally not eligible for enrollment. Only when the mixed histology type is mainly mixed basal cell carcinoma and invasive CSCC is the main histological component, the patients can be enrolled after communication with the investigator and approval.
10. There was at least one measurable lesion (no previous radiotherapy) according to the response evaluation Criteria for solid tumors, version 1.1 (RECIST V1.1). For nonbody surface lesions, accurate measurement by computed tomography (CT) or magnetic resonance imaging (MRI) (intravenous contrast medium is preferred) at baseline showed a long diameter ≥10 mm (except lymph nodes, whose short axis must be ≥15mm), and the lesions were suitable for repeated accurate measurement; For body surface lesions, calipers are required to accurately measure and show their long diameter ≥10 mm and clear lesion edge for repeated and accurate measurement. If the body surface lesions are deeply invasive lesions, CT or MRI is preferred for accurate measurement by referring to non-body surface lesions. A lesion located in a previously irradiated area clearly demonstrated progression that met the RECIST V1.1 criteria (surface lesions must be confirmed as disease progression by biopsy), then the lesion was considered measurable.
11. The subject shall consent to biopsy of the target lesion when the investigator deems it necessary for pathological confirmation.
12. Previous antitumor therapy was required to meet the following criteria: 1. The interval between systemic radiation therapy and the first dose of the study was ≥3 weeks, and the interval between local radiation therapy or bone metastases was ≥2 weeks. No dose of radiation was taken within 8 weeks before the first dose of this study; 2. The interval between previous chemotherapy and previous targeted therapy and the first administration of this study was ≥4 weeks, or ≥ 5 half-lives of the drug (whichever occurred first); 3. The interval between the first administration of immunotherapy, biologic therapy (tumor vaccine, cytokine or tumour-controlling growth factor), endocrine therapy, tumor embolization or other antitumor therapies including Chinese herbal therapy with antitumor indications was ≥4 weeks;
13. Having full organ and bone marrow function, as defined below:
14. Blood routine: absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count (PLT) ≥90×109/L; Absolute white blood cell count (WBC) ≥3.0×109/L; Hemoglobin content (HGB) ≥90 g/L. Note: It is not recommended to use G-CSF, GM-CSF, red blood cell transfusion, platelet transfusion and other interventions to reach the normal range within 14 days before examination.
15. Liver function: total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN); If TBIL > 1.5×ULN, binding bilirubin ≤ULN; For subjects with liver metastases or a history/suspicion of Gilbert's syndrome (persistent or recurrent hyperbilirubinemia, primarily unbound bilirubin hypertrophy, with no evidence of hemolysis or liver disease). TBIL acuities were 3 x ULN. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5×ULN for subjects without liver metastases; For subjects with liver metastases, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤5×ULN.
16. Renal function: serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance (CCr) ≥50 mL/min; 4) Adequate coagulation function, defined as prothrombin time (PT) and partially activated thrombin time (APTT) ≤1.5× upper limit of normal (ULN); If the subject was receiving anticoagulant therapy, the PT or INR was within the prescribed range for the anticoagulant.
17. Female subjects of childbearing age or male subjects whose sexual partners are women of childbearing age are required to use effective contraception throughout the treatment period and for 6 months after the end of treatment.
18. Signed a voluntary informed consent, understanding of the study and being willing to follow and able to complete all trial procedures.

Exclusion Criteria:

1. Received other immunomodulator therapy within 4 weeks before the first dose of this study, or had an immune-related adverse event of grade 1 or higher within 90 days before the first dose of this study; Or discontinuation of immunomodulator therapy due to toxicity during previous treatment. These immunomodulators include therapeutic vaccines, cytokine therapy, or immune checkpoint related therapies such as anti-CTLA4 and OX-40.
2. Previous antitumor therapy targeting PD-1/PD-L1 signaling pathway;
3. Participating in another interventional clinical study, except participating in an observational (non-interventional) clinical study or being in the follow-up phase of an interventional study;
4. Received any investigational drug within 4 weeks prior to the initial administration of the investigational drug;
5. Use of immunosuppressive drugs within 4 weeks prior to the first administration of the study drug, excluding

1) intranasal inhaled topical steroid treatment or topical steroid injection (e.g., intra-articular injection); 2) Systemic corticosteroid treatment not exceeding 10 mg/ day of prednisone or its equivalent physiological dose;

2) Glucocorticoids as prophylaxis for allergic reactions (e.g. pre-CT)

6. The need for long-term systemic hormone or any other immunosuppressive drug therapy does not include inhaled hormone therapy;

7. Toxicities due to previous antitumor therapy that did not return to NCI CTCAE V5.0 grade 0 or 1 or the level specified by the enrollment criteria (excluding hair loss, fatigue, or grade 2 or less endocrine related adverse events due to radiation therapy) were present 4 weeks before the first administration of the study drug;

8. Receive live attenuated vaccine within 4 weeks prior to the first administration of the study drug or planned during the study period;

9. Had a major surgical procedure (craniotomy, thoracotomy, or laparotomy, or otherwise as defined by the investigator) within 4 weeks prior to the initial administration of the study drug or had an unhealed fracture or was expected to have a major surgery during the duration of the study. Note: Local surgical treatment of isolated lesions is acceptable for palliative care purposes;

10. No radiographic enhanced radiographic assessment could be performed (either iodine-enhanced CT or gadolinium MRI could be enrolled). If other conditions are met, any contrast-enhanced radiography cannot be accepted, but comprehensive tumor evaluation can be performed by caliper measurement, and the study can be enrolled after communication with the investigator.

11. Other antitumor therapy (palliative radiotherapy permitted) is anticipated during the trial treatment;

12. A history of pneumonia requiring hormonal therapy, or interstitial lung disease (including past and present history), with the exception of local interstitial pneumonia due to radiation therapy;

13. Known central nervous system (CNS) metastases and/or spinal cord compression and/or cancerous meningitis,

14. History of pIA. Patients with asymptomatic brain metastases (i.e., no neurologic symptoms, no need for glucocorticoid therapy, and no lesions > 1.5 cm) or stable symptoms after treatment of brain metastases were eligible for participation if they met all of the following criteria:

15. Measurable lesions outside the central nervous system; No mesencephalon, pons, cerebellum, meninges, medulla oblongata or spinal cord metastases; Participants were clinically stable for at least 4 weeks, had no evidence of new or expanded brain metastases, and had stopped corticosteroid and anticonvulsant therapy for at least 14 days prior to study treatment;

16. Active, known or suspected autoimmune disease (see Annex 1) or a history of the disease within the previous 2 years (vitiligo, psoriasis, alopecia or Grave's disease that has not required systematic treatment in the last 2 years, Hypothyroidism requiring only thyroid hormone replacement therapy and type 1 diabetes requiring only insulin replacement therapy were eligible).

17. Acute or chronic active hepatitis B [defined as hepatitis B surface antigen (HbsAg) and/or hepatitis B core antibody (HbcAb) positive and hepatitis B virus (HBV) DNA copy number ≥1×103 copies /ml or ≥200 copies /ml IU/ml] or positive for acute or chronic active hepatitis C (HCV) antibody; Subjects with positive HCV antibody but negative RNA test were allowed to enroll

18. Uncontrolled co-morbidities such as

1. Severe infection occurring within 4 weeks prior to study treatment initiation, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia; Or patients who received therapeutic oral or intravenous antibiotics within 2 weeks before starting study treatment and who received prophylactic antibiotics (e.g., to prevent urinary tract infection or chronic obstructive pulmonary disease) were enrolled;
2. HIV-infected persons (HIV antibody positive);
3. History of myocarditis;
4. Symptomatic congestive heart failure (New York Heart Association Class II-IV) or symptomatic or poorly controlled arrhythmias;
5. uncontrolled arterial hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100 mmHg) despite standard treatment;
6. Had any arterial thromboembolic event, including myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack, in the 6 months prior to enrollment;
7. require immediate intervention of esophageal or gastric varices (binding or hardening treatment, for example) or according to the researchers' opinions or consulting experts of gastroenterology and hepatology experts think the bleeding risk is higher, evidence of the portal hypertension (including imaging examination showed splenomegaly) or a history of varices bleeding of the subjects in the group of the first 3 months must undergo endoscopic evaluation;
8. Any life-threatening bleeding event or grade 3 or 4 gastrointestinal/varicose bleeding event requiring blood transfusion, endoscopic or surgical treatment within 3 months prior to study enrollment;
9. A history of deep vein thrombosis, pulmonary embolism, or any other major thromboembolism in the 3 months prior to enrollment (implantable venous port or catheter origin thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism);
10. Portal vein tumor thrombus involves both the main portal vein and the left and right branches, or the main portal vein, superior mesenteric vein and inferior vena cava tumor thrombus;
11. Uncontrolled metabolic disorders or secondary reactions to other non-malignant organ or systemic diseases or cancers that may lead to higher medical risks and/or uncertainty in survival evaluation;
12. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh > 7 or more severe cirrhosis;
13. Subjects at risk for bowel obstruction or perforation (including but not limited to a history of acute diverticulitis, abdominal abscess, or abdominal cancer) or any of the following: inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea;
14. Significant malnutrition, such as the need for intravenous nutrient supplementation; Malnutrition was not corrected for more than 4 weeks before the first dose of study treatment.
15. Tumor invasion of surrounding important organs (such as mediastinal great vessels, superior vena cava, trachea, esophagus, etc.) or risk of esophagotracheal fistula or esophagopleural fistula.
16. After esophageal or tracheal stent implantation
17. Abnormal values of other acute or chronic diseases or laboratory tests that could increase the risk associated with study participation or study drug administration or interfere with the interpretation of study results and, at the investigator's discretion, classify the subject as ineligible for study participation;
18. or neurological, psychiatric/social conditions that affect compliance with study requirements, significantly increase the risk of adverse events, or affect the subject's ability to provide written informed consent.

19. A known history of primary immunodeficiency;

20. Known active tuberculosis or active syphilis;

21. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;

22. Patients who had a history of gastrointestinal perforation and/or fistula within 6 months prior to study enrollment and were not cured by surgery;

23. Accompanied by uncontrolled third space effusion requiring repeated drainage, such as pleural effusion, ascites, pericardial effusion, etc. (patients who do not need drainage effusion or have no significant increase in effusion within 3 days after stopping drainage can be enrolled);

24. Patients who had developed other malignancies in the 5 years prior to enrollment, except for cured cervical carcinoma in situ/cutaneous basal cell carcinoma/breast ductal carcinoma in situ and radical prostate cancer with no detectable prostate-specific antigen (PSA) for at least 3 years;

25. The subject is known to have had a previous severe allergic reaction to other monoclonal antibodies or to any of the study drug preparation components; Pregnant or lactating female subjects.

26.Patients with comorbidities that, in the judgment of the investigator, seriously endanger the safety of the patients or interfere with the completion of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to approximately 24months
  From initiation of treatment to progression of the disease
Overall survival | Up to approximately 120months
  Time from the start of treatment to death

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No